CLINICAL TRIAL: NCT01778439
Title: A Phase 1 Dose Escalation Study of OMP-52M51 in Subjects With Solid Tumors
Brief Title: A Dose Escalation Study of OMP-52M51 in Subjects With Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: OncoMed Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Organization: Mereo BioPharma (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 52M51-002
Record Dates: First submitted 2013-01-24; First posted 2013-01-29 (Estimated); Last update posted 2020-08-11 (Actual); Status verified 2020-08

CONDITIONS: Relapsed or Refractory Solid Tumors
Keywords: Phase 1; Dose escalation; relapsed or refractory; solid tumor
MeSH Terms: conditions — Recurrence

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- OMP-52M51 (Experimental)
  Interventions: Drug: OMP-52M51

INTERVENTIONS:
Drug: OMP-52M51

SUMMARY:
This is an open-label Phase 1a dose escalation study of single-agent OMP-52M51 in subjects with relapsed or refractory solid tumors. Study includes a dose escalation phase and expansion phase. Subjects will be assessed for safety, immunogenicity, pharmacokinetics, biomarkers, and efficacy.

ELIGIBILITY:
Inclusion Criteria:

Subjects must meet all of the following criteria to be eligible for the study:

1. Age >18 years
2. ECOG performance status <2 (see Appendix B)
3. Solid tumor malignancy for which there is no remaining standard therapy or either refuse or are not considered to be candidates for any remaining standard therapy.
4. Must have a tumor that is measurable or evaluable per RECIST v1.1 in the dose escalation phase. In the expansion cohort(s), subjects must have measurable disease.
5. Subjects must have Formalin-Fixed, Paraffin-Embedded (FFPE) tissue available either archived or fresh core or punch needle biopsied at study entry (two fresh cores/punches preferred whenever possible) for determination of Notch1 pathway activation status.
6. Must have received their last chemotherapy, biologic, radiotherapy, or investigational therapy at least 4 weeks prior to enrollment; 6 weeks if the last regimen included BCNU or mitomycin C.
7. Subjects must have normal organ and marrow function as defined below:

   * Absolute neutrophil count >1500/mL without growth factor support in the past 7 days
   * Platelets >100,000/mL without transfusions in the past 7 days
   * Total bilirubin <1.5 X institutional upper limit of normal (ULN) (<2X ULN for subjects with Gilbert's syndrome)
   * AST (SGOT) and ALT (SGPT) <3 X institutional ULN (for subjects with hepatic involvement <5 X institutional ULN but cannot be associated with elevated bilirubin)
   * PT/INR and aPTT within 1.5 X institutional ULN
   * Creatinine <1.5 X institutional ULN OR
   * Creatinine clearance >60 mL/min/1.73 m2 for subjects with creatinine levels above institutional normal
   * Normal Ejection Fraction (>50%) on ECHO scan or MUGA
8. Women of childbearing potential must have had a prior hysterectomy or have a negative serum pregnancy test and be using adequate contraception prior to study entry and must agree to use adequate contraception from study entry through at least 6 months after discontinuation of study drug. Men must also agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry and from study entry through at least 6 months after discontinuation of study drug. Should a woman enrolled in the study or a female partner of a man enrolled in the study become pregnant or suspect she is pregnant while participating in this study or within 6 months after discontinuation of study, she should inform the Investigator immediately.
9. Ability to understand and the willingness to sign a written informed consent document

Exclusion Criteria:

Subjects who meet any of the following criteria will not be eligible for participation in the study:

1. Currently receiving any therapeutic treatment for their malignancy including other investigational agents
2. Prior treatment with gamma secretase inhibitors or other Notch 1 inhibitors
3. Uncontrolled seizure disorder, active neurologic disease, or active CNS involvement except for individuals who have previously-treated CNS metastases, are asymptomatic, and have no requirement for higher doses of corticosteroids (> prednisone 10mg orally per day) or anti-seizure medication for at least 4 weeks prior to first dose of study drug.
4. History of a Grade 4 allergic reaction attributed to humanized or human monoclonal antibody therapy
5. Significant intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements
6. Pregnant women or nursing women
7. Ongoing malignancies or malignancies in remission <3 years other than the malignancies included in this trial. Patients with history of known squamous cell skin cancers within the past 3 years will not be included in this trial. The following prior malignancies are allowable irrespective of when they occurred: in situ carcinoma of the cervix, in situ ductal breast cancer, and low-grade local bladder cancer.
8. Subjects with known HIV infection
9. Known bleeding disorder or coagulopathy
10. Known endobronchial lesions and/or lesions infiltrating major pulmonary vessels.
11. Hemoptysis in excess of 2.5 mL(or one-half teaspoon) within 8 weeks of first dose of study drug.
12. Subjects receiving heparin, warfarin, or other similar anticoagulants, except for subjects on low molecular weight heparin for DVT/PE prophylaxis. Note: Subjects may be receiving low-dose aspirin and/or non-steroidal anti-inflammatory agents.
13. New York Heart Association Classification II, III, or IV (see Appendix D)
14. Subjects with poorly controlled blood pressure (defined as systolic blood pressure ≥140 mmHg or diastolic blood pressure ≥90 mmHg) that is not responsive to medical therapy. Subjects taking antihypertensive medications must be taking ≤2 medications to obtain this level of blood pressure control.

    NOTE: Initiation or adjustment of antihypertensive medication(s) is permitted prior to study entry.
15. Subjects with ECG evidence of ischemia or ≥Grade 2 ventricular arrhythmia, subjects who have a history of acute myocardial infarction within 6 months, or subjects with unstable angina.
16. Subjects with known clinically significant gastrointestinal disease including, but not limited to:

    * inflammatory bowel disease
    * active peptic ulcer disease
    * known intraluminal metastatic lesion(s) with risk of bleeding
    * history of abdominal fistula, GI perforation, or intra-abdominal abscess within 28 days prior to beginning study treatment
17. Subjects with diarrhea at time of enrollment or have an ongoing requirement for anti diarrheal therapy

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2013-02; Primary Completion 2016-07 (Actual); Study Completion 2016-07 (Actual)

PRIMARY OUTCOMES:
Safety profile of OMP-52M51 in subjects with relapsed or refractory solid tumors | Subjects will be assessed for DLTs from Days 0-29. Adverse events will be reported through 30 days after the last dose

SECONDARY OUTCOMES:
Pharmacokinetics (PK) of OMP-52M51 in subjects with relapsed or refractory solid tumors | PK analyses at various time points following the 1st and 2nd doses, immediately pre and post-dose for all subsequent doses at treatment term, every 4 weeks after discontinuation of study drug or 12 weeks
  Apparent half life, AUC, clearance, volume of distribution
Immunogenicity | Assessed at baseline, prior to each dose, at treatment termination and every 4 weeks after the discontinuation of the study drug for 12 weeks.
Preliminary Efficacy | Evaluation for response will be assessed on day 70 of study and every 8 weeks (or 9 weeks for Q3W schedule) thereafter and will be based on RECIST v1.1.

CONTACTS AND LOCATIONS:
Locations (6):
- United States (6):
  - University of California, San Francisco/Helen Diller Cancer Institute, San Francisco, California
  - University of Colorado Denver -RCI-South Tower, Aurora, Colorado
  - Karmanos Cancer Institute (KCI), Detroit, Michigan
  - Wayne State University/Oncology Karmanos Cancer Institute, Detroit, Michigan
  - The University of Texas MD Anderson Cancer Center, Houston, Texas
  - South Texas Accelerated Research Therapeutics, LLC, San Antonio, Texas

REFERENCES:
- [Derived] Ferrarotto R, Eckhardt G, Patnaik A, LoRusso P, Faoro L, Heymach JV, Kapoun AM, Xu L, Munster P. A phase I dose-escalation and dose-expansion study of brontictuzumab in subjects with selected solid tumors. Ann Oncol. 2018 Jul 1;29(7):1561-1568. doi: 10.1093/annonc/mdy171. PMID 29726923